CLINICAL TRIAL: NCT06585670
Title: Effects of a Digital Mindfulness and Meditation Intervention on Mental Health and Vision-Related Quality of Life in Adults With Non-infectious Uveitis
Brief Title: Mindfulness Approach for Reducing Anxiety and Gloom in Ocular Inflammatory Diseases
Acronym: MARiGOLD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Calm.com, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-38336
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Non-infectious Uveitis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Mindfulness Intervention Arm (Experimental): Participants in the intervention arm will be asked to engage with the digital meditation and mindfulness modules administered through the Calm Health platform for at least 10 minutes per day for 8 weeks.
  Interventions: Other: Calm Health - smartphone application
- Non-Intervention Arm (No Intervention): Participants in the non-intervention arm will not have access to the invite-only Calm Health mobile application for the first 8 weeks of the study. They will be instructed not to use any other digital mindfulness or meditation platform over the course of the study. They will be granted access to the mobile application after 8 weeks since their enrollment have elapsed.

INTERVENTIONS:
Other: Calm Health - smartphone application — Participants randomized to the intervention arm of the study will be given free access to a mobile phone application called Calm Health, which they will use to engage in guided meditation and mindfulness modules for at least 10 minutes per day for 8 weeks.
  Arms: Digital Mindfulness Intervention Arm

SUMMARY:
The proposed study is a block-randomized, controlled trial to evaluate the effects of a digital meditation and mindfulness practice on mental health in patients with non-infectious uveitis.

DETAILED DESCRIPTION:
Non-infectious uveitis is an immune-mediated inflammatory disease of the eye that can occur alone or be associated with other autoimmune diseases. This chronic condition can be isolating and complex for patients to manage, leading to increased rates of anxiety and depression symptoms in uveitis patients compared to the general population.

In collaboration with Calm Health, the investigators aim to evaluate the efficacy of Calm Health's meditation, mindfulness, and clinical programs in reducing symptoms of anxiety and depression, as well as perceived stress, in patients. Overall, the investigators aim to collect data on the value of supplementing medical care with an accessible digital mental health resource.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 or older at time of enrollment.
* Is willing to download Calm Health on their smartphone
* Is able to operate a smartphone & Calm Health without assistance
* Is able to read words on a screen without assistance
* Diagnosis of non-infectious uveitis

Exclusion Criteria:

* Is under 18 at time of enrollment.
* Has started taking a new anti-depressant, anti-anxiety, or other psychiatric medication to improve mood within the past month.
* Plans to start taking a new anti-depressant, anti-anxiety, or other psychiatric medication to improve mood in the next 12 weeks.
* Has started any type of psychotherapy within the past 3 months.
* Plans to start any type of psychotherapy within the next 12 weeks.
* Already has a mindfulness/meditation app on their smartphone.
* Is unable to operate a smartphone or read words on a screen without assistance.
* Is unable or unwilling to download the Calm Health app on their smartphone.
* Does not consent to their anonymized data being collected via Calm Health app.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Anxiety Symptoms | The primary outcome will be measured at 8 weeks.
  The severity of anxiety symptoms of participants will be assessed by the 7-item Generalized Anxiety Disorder (GAD-7) questionnaire, which is a diagnostic self-report scale that can be used to screen for and assess the severity of Generalized Anxiety Disorder (GAD). The questionnaire asks the participant to self-report the frequency of 7 different anxiety symptoms on a scale of 0 (not at all) to 3 (nearly every day) over the past two weeks. Scores ranging from 0-4 represent none to minimal anxiety, scores ranging from 5-9 indicate mild anxiety, scores 10-14 indicate moderate anxiety, and scores ranging from 15-21 indicate severe anxiety. For this study, we are defining a clinically meaningful improvement in anxiety symptoms as a decrease of 2.6 points on the GAD-7, which falls within the range of values referenced in the literature.

SECONDARY OUTCOMES:
Depression Symptoms | This secondary outcome will be measured at 8 weeks.
  The severity of depressive symptoms of participants will be assessed by the 9-item Patient Health Questionnaire (PHQ-9), which is a diagnostic self-report scale that can be used to screen for and assess the severity of depression. The questionnaire asks the participant to self-report the frequency of 9 different depressive symptoms on a scale ranging from 0 ("not at all") to 3 ("nearly every day") over the last two weeks. Total scores ranging from 1- 4 indicate minimal depression, scores ranging from 5-9 indicate mild depression, scores ranging from 10-14 indicate moderate depression, scores 15-19 indicate moderately severe depression, and scores ranging from 20-27 indicate severe depression. A clinically meaningful improvement in symptoms of depression is defined as a decrease of 1.7 points on the PHQ-9.
Perceived Stress | This secondary outcome will be measured at 8 weeks.
  The severity of perceived stress in participants will be assessed by the 10-item Perceived Stress Scale (PSS-10), which is a self-report scale that can be used to evaluate the severity of stress that young people and adults aged 12 and above experience in their daily life, over the past month. The survey asks the participant about feelings related to unpredictability, overwhelm, loss of control, and coping with the pace of everyday life. The survey asks the participant to describe the frequency of these feelings on a scale ranging from 0 ("never") to 4 ("very often"). Higher scores indicate higher stress; scores ranging from 0-13 indicate low stress, scores ranging from 14-26 indicate moderate stress, and scores ranging from 27-40 indicate high perceived stress. A clinically meaningful improvement in perceived stress is defined as a decrease of 11 points on the PSS-10.
Vision-Related Quality of Life | This secondary outcome will be measured at 8 weeks.
  The vision-related quality of life of participants will be assessed by the 25-item National Eye Institute Visual Functioning Questionnaire (NEI VFQ-25), which measures the dimensions of self-reported vision-targeted health status that are most important for patients who have chronic eye diseases. The survey is designed to measure the influence of visual disability and visual symptoms on emotional well-being, social functioning, and daily visual functioning. Scores range from 0-100, with higher scores representing a higher vision-related quality of life. A clinically meaningful improvement in vision-related quality of life is defined as increase of 14 points on the NEI VFQ-25.

OTHER OUTCOMES:
Adherence-Based Subgroup Analyses | Levels of adherence will be determined at the end of their 8-week study period.
  Prespecified subgroup analyses for primary and secondary outcomes will examine the difference in mean GAD-7, PHQ-9, PSS-10, and VFQ-25 score changes between control and intervention participants at the prespecified levels of adherence:
  1. Completed the required 10-minute app usage requirement for 1a) 75%, 1b) 50%, or 1c) 25% of the days within the 8-week study period.
  2. Completed any minutes of app usage for 2a) 75%, 2b) 50%, or 2c) 25% of the days within the 8-week study period.
  An additional analysis will examine the difference in mean GAD-7, PHQ-9, PSS-10, and VFQ-25 score changes between control and intervention participants, while adjusting for total minutes of app usage over the study period as a continuous variable.

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Acharya, MD, MS, Principal Investigator — UCSF, Proctor Foundation
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen KD, Paniagua SM, Kazanis W, Jones S, Potter JS. Quality of life among women diagnosed with breast Cancer: A randomized waitlist controlled trial of commercially available mobile app-delivered mindfulness training. Psychooncology. 2018 Aug;27(8):2023-2030. doi: 10.1002/pon.4764. Epub 2018 Jun 1. PMID 29766596
- [Background] Niemeyer KM, Gonzales JA, Doan T, Browne EN, Rao MM, Acharya NR. Time Trade-off Utility Values in Noninfectious Uveitis. Am J Ophthalmol. 2019 Dec;208:47-55. doi: 10.1016/j.ajo.2019.06.005. Epub 2019 Jun 13. PMID 31201795